CLINICAL TRIAL: NCT02857400
Title: Evaluation of an Organized Consultation "Return Home" of Patients With a Cancer (CREDO)
Acronym: CREDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16GENE11
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: METASTATIC CANCER
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (standard) (Other)
  Interventions: Other: current standard of care
- Arm B (experimental) (Experimental)
  Interventions: Other: CREDO standard of care

INTERVENTIONS:
Other: current standard of care — connection documentation faxed to GP (General practitioner) on the day of patient's discharge
  Arms: Arm A (standard)
Other: CREDO standard of care — organized consultation "return home" between patient, GP DESC (diploma of complementary specialized study) and patient's referent GP
  Arms: Arm B (experimental)

SUMMARY:
Prospective, open label, randomized and multicentric study evaluating the efficacy of an organized consultation "return home" compared to a current standard of care in patient hospitalized due to metastatic solid tumor cancer.

Subject will be randomized (1:1) as described below :

• Arm A (standard) : current standard of care ; connection documentation faxed to GP ( General practitioner) on the day of patient's discharge Arm B (experimental) : CREDO standard of care, organized consultation "return home" between patient, GP DESC (diploma of complementary specialized study) and patient's referent GP

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 years old
2. Subject hospitalized in an oncology dedicated center for administration of the first chemotherapy cycle.
3. Subject with metastatic solid tumor whatever the organ
4. subject planned to be discharged home after chemotherapy administration
5. Affiliated to the French social security system.
6. Subjects must provide written informed consent prior to any study-specific procedure or assessment

Exclusion Criteria:

1. Subject included in another trial evaluating the pathways care
2. Pregnant or breastfeedings women
3. Subject law protected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of an organized consultation "return home" of patients with a metastatic cancer | up to 12 months
  Evaluation of number of non planned consultation and hospitalization compared to current standard of care

SECONDARY OUTCOMES:
Comparison of the 2 standard of care (current and CREDO) regarding subject' satisfaction | up to 12 months
  phone call , specific question
Comparison of the 2 standard of care (current and CREDO) regarding subject's quality of life | up to 12 months
  quality of life questionnaire
Identification of the conformity of the standard of care regarding the place of care | up to 12 months
  Comparison with the initial predefined place of standard of care
To quantify the caregiver burden in the 2 standard of care (current and CREDO) | up to 12 months
  Zarit Burden Interview
To assess the medical and economic consequences of the 2 standard of care (current and CREDO) | up to 12 months
  A cost effectiveness analysis will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eve ROUGE BUGAT, MD, Principal Investigator — Institut Claudius Regaud
Locations (3):
- France (3):
  - Centre Hospitalier Auch, Auch
  - Hopital Rangueil, Toulouse
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gimenez L, Grosclaude P, Druel V, Costa N, Delpierre C, Molinier L, Delord JP, Rouge Bugat ME. Study protocol of the CREDO randomised controlled trial: evaluation of a structured return home consultation for patients suffering from metastaticcancer. BMJ Open. 2023 Jan 30;13(1):e062219. doi: 10.1136/bmjopen-2022-062219. PMID 36717134